CLINICAL TRIAL: NCT05519683
Title: Effects of Home-based TEA for Abdominal Pain in Patients With Irritable Bowel Syndrome (IBS)
Brief Title: Home Transcutaneous Electrical Acustimulation (TEA)
Acronym: Home-TEA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Borko Nojkov, Assistant Professor - Specialty Gastroenterology, Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00217301; 5UH3NS115108-04 (NIH)
Record Dates: First submitted 2022-08-18; First posted 2022-08-29 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-08

CONDITIONS: Irritable Bowel Syndrome With Constipation
Keywords: Irritable Bowel Syndrome with Constipation; Constipation; Irritable Bowel Syndrome; Colon, Irritable; Irritable Colon
MeSH Terms: conditions — Constipation; Irritable Bowel Syndrome | interventions — Escitalopram

STUDY DESIGN:
Masking Description: One quarter of participants will be in each arm. Those randomized to device arms will not be informed of their parameters. Those in the drug arm will be informed of their arm soon after randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- TEA at location A (Experimental): The TEA device administers a mild electrical shock through the skin, similar to acupuncture. Stimulation will be performed twice daily, morning and evening for 45 minutes for 8 weeks. Location sets are described in the protocol, which will be shared with results reporting but are not provided here to maintain masking and, therefore, to safeguard scientific integrity.
  Interventions: Device: TEA
- TEA at location B (Sham Comparator): The TEA device administers a mild electrical shock through the skin, similar to acupuncture. Stimulation will be performed twice daily, morning and evening for 45 minutes for 8 weeks. Location sets are described in the protocol, which will be shared with results reporting but are not provided here to maintain masking and, therefore, to safeguard scientific integrity.
  Interventions: Device: TEA
- TEA at location C (Experimental): The TEA device administers a mild electrical shock through the skin, similar to acupuncture. Stimulation will be performed twice daily, morning and evening for 45 minutes for 8 weeks. Location sets are described in the protocol, which will be shared with results reporting but are not provided here to maintain masking and, therefore, to safeguard scientific integrity.
  Interventions: Device: TEA
- Escitalopram treatment (Experimental): This arm will receive treatment with the chemical neuromodulator escitalopram (Lexapro) at 10 mg once per day for 8 weeks. Lexapro is often used as a standard treatment for IBS.
  Interventions: Drug: Lexapro

INTERVENTIONS:
Device: TEA — The TEA device administers a mild electrical shock through the skin, similar to acupuncture. Location sets are described in the protocol, which will be shared with results reporting but are not provided here to maintain masking and, therefore, to safeguard scientific integrity.
  Other Names: Transcutaneous Electrical Acustimulation
  Arms: TEA at location A; TEA at location B; TEA at location C
Drug: Lexapro — This arm will receive treatment with the chemical neuromodulator escitalopram (Lexapro) at 10 mg once per day for 8 weeks. Lexapro is often used as a standard treatment for IBS.
  Other Names: escitalopram
  Arms: Escitalopram treatment

SUMMARY:
This study will assess the efficacy of two active treatments with TEA and a chemical neuromodulator (escitalopram aka Lexapro) versus a sham comparator or control group on abdominal pain.

DETAILED DESCRIPTION:
The aim of this study is to investigate the potential of TEA to treat abdominal pain in participants with IBS with constipation (IBS-C). The study also aims to compare the electrical neuromodulation therapy (TEA) with medical neuromodulation therapy (escitalopram) in their ability to treat abdominal pain and improve the autonomic dysfunction in participants with IBS-C. This project will investigate the impact of 3 active treatment interventions vs. a sham control intervention on abdominal pain and other IBS symptoms in participants with IBS-C. This is a parallel-group study in which the participants will be divided into 4 treatment groups designed to investigate the feasibility of TEA using optimized parameters in comparison with medical neuromodulation therapy (escitalopram) and sham-TEA. The treatment will be home-based and last for a period of 8 weeks. To preserve scientific integrity and effective masking, certain details of arms and interventions will be made more precise upon or prior to reporting results

ELIGIBILITY:
Inclusion Criteria:

* Those with ongoing and symptomatic Irritable Bowel Syndrome with Constipation (IBS-C)
* Significant mean worst abdominal pain severity (as defined by the study protocol, which will be shared with results reporting) on a Visual Analog Scale (VAS) pain score during the Phase-in period
* Symptoms present at least 1 day/week in the last 3 months with symptom onset at least 6 months prior to the diagnosis.
* Abdominal pain is not adequately relieved at the time of screening and the time of randomization.

Exclusion Criteria:

* Unrelated active disorder which may involve abdominal pain, such as inflammatory bowel disease, diabetes or unstable thyroid disease.
* Pregnancy, plans to become pregnant, or lactation. Any potential patient of child-bearing potential will complete a pregnancy test at Visit 1 and if the test is positive that individual will be excluded from future participation.
* Any other condition, which in the opinion of the investigator would impede compliance or hinder the completion of the study
* A history of abdominal surgery (other than cholecystectomy or appendectomy)
* Active use of prucalopride, domperidone, alosetron, tegaserod, warfarin, antipsychotic (e.g., Seroquel, Risperdal), antidiarrheal, or frequent (>2 days/week) use of opioid or antispasmodic medication. Those who frequently use Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) will also be excluded.
* Ongoing use of Selective Serotonin Reuptake Inhibitors (SSRIs), Serotonin and Norepinephrine Reuptake Inhibitors (SNRIs), or any other serotonin-active medications, including tricyclic antidepressants (TCAs). Individuals on chronic SSRI therapy, including escitalopram, at the initial evaluation will not be enrolled in the study.
* Inability to avoid the following medications: tricyclic antidepressants, Monoamine Oxidase (MAO) inhibitors including, intravenous methylene blue, linezolid, and pimozide, as well as triptans, fentanyl, lithium, tramadol, tryptophan, buspirone, amphetamines, and St. John's Wort. - - Participants will be informed that MAO inhibitors cannot be used within 14 days of starting or stopping escitalopram.
* Known hypersensitivity to escitalopram or citalopram including any of the inactive ingredients of these formulations.
* Known allergy to adhesive Electrocardiogram (ECG) electrodes.
* Known angle-closure glaucoma, bipolar disorder, history of seizures or prior suicide attempt or known suicidal thoughts.
* Known QTc prolongation or receiving scheduled therapy with a medication associated with prolongation of QTc (screening to be completed at recruitment as detailed above).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in abdominal pain/discomfort via daily Visual Analog Scale (VAS) survey | Daily for 14 weeks
  Participants will complete a daily VAS survey to measure daily discomfort. There are four metrics measured in this form, abdominal pain, abdominal bloating, abdominal fullness, and abdominal cramping. These are scored on a line from 0 to 10, with 0 being the lowest (no pain) and 10 being the highest (worst imaginable pain)
  These scores will be totaled each day and compared from day 0 to day 98, or the end of week 14.
Change in global abdominal pain | Weekly for 14 weeks
  Participants will complete a weekly VAS survey to monitor for change in discomfort for the week prior when compared to prior to starting the study. This contains two questions which ask yes/no questions asking about improvement over the prior week, and one question asking for satisfaction of improvement from 0 to 5, 0 being the lowest (not satisfied) and 5 being the highest (very satisfied).
  These answers will be compared from week 1 to week 14.

SECONDARY OUTCOMES:
Change in quality of life via Irritable Bowel Syndrome - Quality of Life (IBS-QOL) survey | Weekly for 14 weeks
  A self-report quality-of-life measure specific to Irritable Bowel Syndrome (IBS) that can be used to assess the impact of IBS and its treatment. This survey is 34 questions, all scored from 1 to 5, with 1 being the lowest (not at all) and 5 being the highest (a great deal, or extremely). The individual responses to the 34 items are summed and averaged for a total score.
  These answers will be compared from week 0 to week 14
Change in Hospital Anxiety and Depression Scale (HADS) - Anxiety | Weekly for 14 weeks
  Determines levels of anxiety that a person is experiencing by asking 7 questions scored from 0-3, with 0 being the lowest (not at all) and 3 being the highest (most of the time). Responses for each category will be totaled and compared against the below ranges.
  0-7 = normal 8-10 = borderline abnormal 11-21 = abnormal
  Scores will be compared from week 0 to week 14
Change in Hospital Anxiety and Depression Scale (HADS) - Depression | Weekly for 14 weeks
  Determines levels of depression that a person is experiencing by asking 7 questions scored from 0-3, with 0 being the lowest (not at all) and 3 being the highest (most of the time). Responses for each category will be totaled and compared against the below ranges.
  0-7 = normal 8-10 = borderline abnormal 11-21 = abnormal
  Scores will be compared from week 0 to week 14
Change in IBS - Symptom Severity Score (IBS-SSS) | Once every 10 days for 14 weeks
  A survey designed to record and monitor the severity of IBS. The maximum achievable score was 500. Mild, moderate and severe cases were indicated by scores of 75 to 175, 175 to 300 and > 300 respectively.
  Scores will be compared from day 10 to day 90
Daily Stool Diary - Change in number of bowel movements | Daily for 14 weeks
  The Daily Stool Diary will ask how many bowel movements have occurred in the past 24 hours. This will also ask to indicate the number of spontaneous bowel movements (a bowel movement which occurs without use of rescue medications or maneuvers) and number of complete spontaneous bowel movements (a bowel movement which is associated with a feeling of complete evacuation)
  The change in the mean daily number of bowel movements will be averaged over 1 week and compared between the phase-in period and the final week of the treatment period.
Daily Stool Diary - Change in Bristol Stool Form Scale (BSFS) | Daily for 14 weeks
  The Daily Stool Diary will use the BSFS to evaluate the stool consistency for each of the bowel movements in the past 24 hours. The BSFS is scored from 1 to 7, which are defined as follows:
  BSFS Type 1: Separate hard lumps, like nuts BSFS Type 2: Sausage-shaped but lumpy BSFS Type 3: Like a sausage but with cracks on its surface BSFS Type 4: Like a sausage or snake, smooth and soft BSFS Type 5: Soft blobs with clear-cut edges BSFS Type 6: Fluffy pieces with ragged edges, a mushy stool BSFS Type 7: watery, no solid pieces, entirely liquid
  The change in the mean daily scores for Bristol Stool Form Scale will be averaged over 1 week and compared between the phase-in period and the final week of the treatment period.
Daily Stool Diary - Change in abdominal bloating | Daily for 14 weeks
  The Daily Stool Diary will rate the severity of participants abdominal bloating over past 24 hours on a visual analog scale for bloating (0-10 scale), with 0 being the lowest (no bloating) and 10 being the highest (worst imaginable bloating)
  The change in the mean daily scores for abdominal bloating will be averaged over 1 week and compared between the phase-in period and the final week of the treatment period.
Daily Stool Diary - Change sense of urgency | Daily for 14 weeks
  The Daily Stool Diary will assess the sense of urgency with the following question: "Have you felt or experienced a sense of urgency today?" which will be answered with a yes or no.
  The change in the most frequent daily scores for sense of urgency will be calculated over 1 week and compared between the phase-in period and the final week of the treatment period.
Change in Bowel Habits Per Separate IBS-SSS Survey | Once every 10 days for 14 weeks
  This survey (a part of the IBS-SSS which is not factored into the scoring) contains 9 questions asking about bowel habits. This will question the minimum and maximum number of bowel movements per day/week/month, typical location of pain, the effect of IBS pain on work habits.
  Responses will be compared from day 10 to day 90

CONTACTS AND LOCATIONS:
Overall Officials: Borko Nojkov, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be shared. However, the study protocol and the study results will be shared

REFERENCES:
- [Background] Ma D, Han JS, Diao QH, Deng GF, Ping XJ, Jin WJ, Wu LZ, Cui CL, Li XD. Transcutaneous electrical acupoint stimulation for the treatment of withdrawal syndrome in heroin addicts. Pain Med. 2015 May;16(5):839-48. doi: 10.1111/pme.12738. PMID 25989154
- [Background] Jiang Y, Liu J, Liu J, Han J, Wang X, Cui C. Cerebral blood flow-based evidence for mechanisms of low- versus high-frequency transcutaneous electric acupoint stimulation analgesia: a perfusion fMRI study in humans. Neuroscience. 2014 May 30;268:180-93. doi: 10.1016/j.neuroscience.2014.03.019. Epub 2014 Mar 20. PMID 24657460
- [Background] Qu F, Wang FF, Wu Y, Zhou J, Robinson N, Hardiman PJ, Pan JX, He YJ, Zhu YH, Wang HZ, Ye XQ, He KL, Cui L, Zhao HL, Ye YH. Transcutaneous Electrical Acupoint Stimulation Improves the Outcomes of In Vitro Fertilization: A Prospective, Randomized and Controlled Study. Explore (NY). 2017 Sep-Oct;13(5):306-312. doi: 10.1016/j.explore.2017.06.004. Epub 2017 Jun 30. PMID 28915981
- [Background] Yu Y, Wei R, Liu Z, Xu J, Xu C, Chen JDZ. Ameliorating Effects of Transcutaneous Electrical Acustimulation Combined With Deep Breathing Training on Refractory Gastroesophageal Reflux Disease Mediated via the Autonomic Pathway. Neuromodulation. 2019 Aug;22(6):751-757. doi: 10.1111/ner.13021. Epub 2019 Jul 26. PMID 31347247
- [Background] Zhang B, Xu F, Hu P, Zhang M, Tong K, Ma G, Xu Y, Zhu L, Chen JDZ. Needleless Transcutaneous Electrical Acustimulation: A Pilot Study Evaluating Improvement in Post-Operative Recovery. Am J Gastroenterol. 2018 Jul;113(7):1026-1035. doi: 10.1038/s41395-018-0156-y. Epub 2018 Jun 21. PMID 29925916